CLINICAL TRIAL: NCT03363620
Title: Comparison of Arch Expansion Changes Between Passive Self-ligating and Conventional Brackets With Broad Arches After Alignment and Levelling With the Same Arch Protocol: A Randomized Controlled Trial
Brief Title: Comparison of Arch Expansion Changes Between Passive Self-ligating and Conventional Brackets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, ANGELA MARIA SIERRA ANGEL, ORTHODONTIST, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CES101
Record Dates: First submitted 2017-11-04; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Orthodontic Appliance Complication
Keywords: maxillary expansion; self ligating; arch form
MeSH Terms: interventions — Orthodontic Brackets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self ligation brackets damon ormco® (Experimental): the self ligation bracket (damon system) in the orthodontic treatment, was used in the experimental group with the recommended protocol damon arches sequence.
  Interventions: Device: Orthodontic Brackets
- conventional brackets orthos ormco® (Active Comparator): the conventional bracket (orthos system) in the orthodontic treatment, was used in the active comparator group with the recommended protocol damon arches sequence as used in the experimental group.
  Interventions: Device: Orthodontic Brackets

INTERVENTIONS:
Device: Orthodontic Brackets — arch form development in the orthodontic treatment with 2 different kind of ligation brackets with the same arches protocol in the leveling and alignment phase
  Other Names: self ligation brackets
  Arms: self ligation brackets damon ormco®
Device: Orthodontic Brackets — arch form development in the orthodontic treatment with 2 different kind of ligation brackets with the same arches protocol in the leveling and alignment phase
  Other Names: conventional brackets
  Arms: conventional brackets orthos ormco®

SUMMARY:
The purpose of this randomized controlled clinical trial was to compare the transverse development of the arches and the incisor inclination comparing two different ligating systems (SL vs CL) with the same arch form protocol (Damon arch form) and the same disarticulation protocols after the alignment and leveling period of non-extraction patients.

DETAILED DESCRIPTION:
Materials and Methods: Fifty-four subjects were randomly with an electronic randomization program allocated to treatment with either a self-ligating bracket system (Damon Q-slot 0.022", Ormco Corp,) or a conventional bracket system (Orthos-slot 0.022", Ormco Corp). All patients were treated following the same protocol and arch wire sequence: 0.014-inch, 0.018-inch and 0.014x0.025-inch Damon copper nickel-titanium arch wires (Cu-NiTi; Ormco). Lateral cephalograms and study models, taken at prior to treatment (T0) and after alignment and levelling (T1), were used to compare the amount of arch expansion and incisor angulation changes that took place. In the analysis of results in a single observer analyzes the data blindly without knowing which group the patients belonged. Results: Models and cephalograms of the patients and both stages(T0-T1) were measured at the data were analyzed in STATA S.E. Treatment produce statistically significant increases in transverse arch dimensions especially in premolars maxillary (2.8-4.3mm) and mandibullary (2.0-4.2mm) of both group. The expansion in the maxillary arch was similar for both groups, but in the mandibular arch was greater in the self ligation group in about 2 mm more. Conclusions: The treatment with self ligation brackets produced more expansion in the mandibular arch than the conventional ligation brackets when used the same arch Damon protocols.

ELIGIBILITY:
Inclusion Criteria:

1. ANB angle between 0º- 5º
2. Systemically and periodontally healthy subjects not taking any medications.
3. Maxillary and/or mandibular irregularity index (canine-to-canine) between mild to moderate
4. A non-extraction treatment approach.
5. Permanent dentition with second molars erupted or in a functional eruptive phase.

Exclusion Criteria:

1. Systemically and periodontally compromise subjects and taking any medications. (2 ) subjects who did not want participate in the investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
transverse development of the arches | 2 years
  The maxillary and mandibular widths were measured between the cusp tips of the canines, the buccal cusp tips of the first and second premolars and the mesio-buccal cusp tips of the first molars . They were measured using a digital caliper (Starrett 799A-6/150 Digital Caliper, Athol, Massachusetts, USA) positioned parallel to the occlusal plane.

SECONDARY OUTCOMES:
incisor inclination | 2 years
  incisor inclination , the maxillary incisors were measured in the lateral cephalogram, relative to the cranial base (U1-SN) and the palatal plane (U1-PP); the mandibular incisor were related to the mandibular plane (L1/Go-Gn) and NB (L1-NB).

REFERENCES:
- [Background] Atik E, Akarsu-Guven B, Kocadereli I, Ciger S. Evaluation of maxillary arch dimensional and inclination changes with self-ligating and conventional brackets using broad archwires. Am J Orthod Dentofacial Orthop. 2016 Jun;149(6):830-7. doi: 10.1016/j.ajodo.2015.11.024. PMID 27241993
- [Result] Fleming PS, Lee RT, Marinho V, Johal A. Comparison of maxillary arch dimensional changes with passive and active self-ligation and conventional brackets in the permanent dentition: a multicenter, randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):185-93. doi: 10.1016/j.ajodo.2013.03.012. PMID 23910199